CLINICAL TRIAL: NCT04254042
Title: Rationale and Design of a Simple Randomized Trial Evaluating Comparative Effects of Perindopril and Zofenopril in Blacks Hypertensive Patients: Short Term Effects on Cardiac and Oxidative Status With Perindopril or Zofenopril (PEZO-HP) Trial
Brief Title: Comparative Effects of Perindopril and Zofenopril on Blood Pressure Control and Oxidative Status Blacks Hypertensive Patients.
Acronym: PEZO-HP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Responsible Party: Principal Investigator, CN NGANOU-GNINDJIO, MD, MSc, Dr, Principal investigator, Yaounde Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEZO-HP study
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Hypertension
Keywords: Angiotensin Converting Enzymes Inhibitor; Angiotensin II Receptor Blockers; Blood pressure; Oxidative status
MeSH Terms: conditions — Hypertension | interventions — Viacoram; Perindopril; zofenopril

STUDY DESIGN:
Intervention Model Description: PEZO-HP trial is a double blind, randomized, controlled parallel clinical trial conducted at the Yaounde central hospital, Cameroon
Who Masked: Participant, Investigator
Masking Description: The double-blind model is applied to the study. Only the adjudicator, responsible for the distribution of medication knew the different regimes. Perindopril and Zofenopril were packaged in boxes of identical appearance and labeled for each participant by name and number of the randomization program. The randomization and packaging of the drugs was done by an investigator who had no clinical involvement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perindopril Arm (Active Comparator): 10 mg Perindopril tablet per day at 8am (+/- 1 hour) was add to the usual treatment for each patient. Patients are followed-up for a period of 08 weeks.
  Interventions: Drug: Perindopril Arginine
- Zofenopril Arm (Active Comparator): 30 mg Zofenopril tablet per day at 8am (+/- 1 hour) was add to the usual treatment for each patient. Patients are followed-up for a period of 08 weeks.
  Interventions: Drug: Zofenopril, Calcium Salt, (1(R*),2Alpha,4Alpha)-isomer

INTERVENTIONS:
Drug: Perindopril Arginine — 10 mg Perindopril tablet / day will be added to the usual treatment for each patient for a period of 8 weeks.
  Other Names: Perindopril
  Arms: Perindopril Arm
Drug: Zofenopril, Calcium Salt, (1(R*),2Alpha,4Alpha)-isomer — 30 mg Zofenopril tablet / day will be added to the usual treatment for each patient for a period of 8 weeks.
  Other Names: Zofenopril
  Arms: Zofenopril Arm

SUMMARY:
The aim of the study is to compare the short term effect of perindopril and zofenopril in the management of hypertension and the oxydative stress in blacks hypertensive patients.

PEZO-HP is a double-arm, double-blind, randomized and parallel clinical trial conducted at the Yaoundé Central Hospital.

DETAILED DESCRIPTION:
Aim: to determine and compare the short term effect of angiotensin converting in the management of hypertension as well as the oxidative effect of Zofenopril and perindopril in blacks hypertensive patients in the Yaoundé Central Hospital.

Method: A double-arm, double-blind, randomized and parallel clinical trial conducted at the Yaoundé Central Hospital. Hypertensive patients who are not taking angiotensin-converting enzyme inhibitor or angiotensin receptors blockers, are randomize into 2 groups. Depending on the group, the intervention consisted of the administration of Perindopril 10 mg daily or Zofenopril 30 mg daily for 08 weeks. The endpoints were the nycthemeral blood pressure profile, pro oxidant marker (malondialdehyde) and anti-oxidant marker (Ferric reducing antioxidant).

Progress: Recruitment for PEZO-HP was completed in May 2019 with 24 patients.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients
* On a stable atihypertensive therapies (determined by the investigator) for at least 3 months with no classes changes. The pharmacological treatment should not include an angiotensin-converting enzyme inhibitor or angiotensin II receptor blocker
* Subject must not present any contraindication to exercise
* Before any study-specific procedure, the appropriate written informed consent must be obtained.

Exclusion Criteria:

* Side effects affecting life quality of patients (determined by the Data Safety Monitoring Board).
* Withdrawal of consent

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change in nycthemeral blood pressure profile (mmHg) | 8 weeks
  Change in nycthemeral blood pressure profile from baseline to week 08. By using Arterial Blood Pressure Monitoring.

SECONDARY OUTCOMES:
Change in serum concentration of oxidant marker: malondialdehyde (micromol/l) | 8 weeks
  Change in concentration of oxidant marker from baseline to week 8. By spectrophotometer
Change in serum concentration of anti-oxidant markers: Ferric reducing antioxidant Power (micromol) | 8 weeks
  Change in concentration of anti oxidant marker from baseline to week 8. By spectrophotometer

CONTACTS AND LOCATIONS:
Locations (1):
- Yaounde Central Hospital, Cardiology department, Yaoundé, Cameroon